CLINICAL TRIAL: NCT05946408
Title: Effects Of Supervised Antenatal Exercises On Low Back Pain And Depression In Primigravida
Brief Title: Effects of Antenatal Exercises in Primagravida
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01546
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Pregnancy Related
Keywords: Pregnancy Related; antenatal depression; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Prenatal Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Antenatal Exercises (Experimental): Supervised antenatal exercises twice a week an antenatal education
  Interventions: Other: Supervised antenatal exercises
- Antenatal Education (Active Comparator): Antenatal education only
  Interventions: Other: Antenatal Education

INTERVENTIONS:
Other: Supervised antenatal exercises — Supervised antenatal exercises along with education twice a week. Protocol consists of warm up (10 min), Aerobic training (20 mins, 60-75% of max. HR), Strength training (25 minutes), followed by a cool down of 15 minutes.
  The Interventions to be provided for a period of 12 weeks.
  Arms: Supervised Antenatal Exercises
Other: Antenatal Education — Antenatal education at 12th week of pregnancy. Which consists of education on Posture in pregnancy, Role of pelvic floor muscles, Labor and breathing and relaxation techniques.
  Arms: Antenatal Education

SUMMARY:
The goal of this Randomized control trial is to determine the effects of antenatal exercises on low back pain in Primagravida. The main questions it aims to answer are whether supervised antenatal exercises have an effect on low back pain and depression in primagravida.

DETAILED DESCRIPTION:
Females usually tend to avoid physical activity during pregnancy. Concept of antenatal exercises and its effects on low back pain or antenatal depression is yet not common amongst pregnant females in Pakistan. Low back pain and antenatal depression are common in pregnancy. These can have an impact on both their own health and the health of their unborn child. Understanding the benefits of antenatal exercises will encourage pregnant females to engage in regular physical activity. The results of this study will help physical therapists to implement effective exercise interventions for this population.

ELIGIBILITY:
Inclusion Criteria:

* Primagravida
* Single pregnancy
* Diagnosed for risk of Prenatal depression on EDPS >10
* Pregnancy related Low back pain score of 3 to 8 on NPRS for at least 2 weeks.
* Females in 2nd Trimester of pregnancy

Exclusion Criteria:

* Any present or previous pelvic floor dysfunctions diagnosed by health professionals.
* Any physical disability causing inability to perform physical exercises.
* Any contraindications to physical activity according to ACOG
* Pelvic girdle pain (Anterior: Pubic symphysis, Posterior: SI joint Pain, Gluteal Pain, Piriformis syndrome).
* Rheumatoid disorders.
* Low back pain with radiation
* Not engaged in regular exercise.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Low back pain | 12th Week
  Changes from baseline low back pain will be assessed on Numeric pain rating scale. The scale ranges from 0 for no pain to 10 for worse pain.
The Roland Morris Low Back Pain and Disability Questionnaire | 12th Week
  Changes from baseline low back pain related disability will be assessed using Roland Morris low back pain and disability questionnaire. It is a self-report questionnaire consisting of 24 questions that are scored on a dichotomous scale (yes/no). The total score ranges from 0 to 24, with higher scores indicating greater disability.
Beck depression inventory | 12th week
  Changes from baseline antenatal depression will be assessed using Beck depression inventory. A total score of 0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression. Higher total scores indicate more severe depressive symptoms

SECONDARY OUTCOMES:
Multidimensional Fatigue Inventory | 12th week
  Changes from baseline fatigue will be assessed using Multidimensional Fatigue Inventory. The MFI is a 20-item scale designed to evaluate five dimensions of fatigue:
  general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Items are scored on a scale of 1 to 5. For the total score, a higher score represent greater fatigue.
Fear of Childbirth Questionnaire | 12th week
  Changes from baseline The Fear of Childbirth Questionnaire (FCQ) this is 20 item questionnaires for women who are pregnant. Items are scored on a scale of 1 to 5. A higher score indicates greater fear

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ehsan, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Khyber Teaching Hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No